CLINICAL TRIAL: NCT05592743
Title: The Expanded Access Use of Vorasidenib in Patients With IDH1 or IDH2 Mutated Glioma
Brief Title: Vorasidenib Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: Servier (Industry)
Collaborators: Servier Pharmaceuticals, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: VORA-EAP
Record Dates: First submitted 2022-10-19; First posted 2022-10-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Glioma; Recurrence; Disease Attributes; Pathologic Processes; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue
Keywords: Vorasidenib; AG-881; S95032; Glioma; Oligodendroglioma; Astrocytoma; IDH-1; IDH-2
MeSH Terms: conditions — Glioma; Recurrence; Disease Attributes; Pathologic Processes; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Oligodendroglioma; Astrocytoma | interventions — vorasidenib

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Vorasidenib — Oral therapy
  Other Names: AG-881, S95032

SUMMARY:
This is an expanded access program to provide vorasidenib for treatment of patients 12 years or older with IDH1- or IDH2-mutated glioma.

DETAILED DESCRIPTION:
This expanded access program is designed to provide access to vorasidenib for patients with IDH1- or IDH2-mutated glioma who are not eligible for other vorasidenib clinical trials, and who in the opinion of the treating oncologist would potentially benefit from treatment with vorasidenib.

Safety assessments (including vital signs, hematology, and serum chemistry) occur every two weeks for the first two cycles (28 day each cycle), then monthly for the duration of treatment. Treatment with vorasidenib will continue until, in the clinical judgement of the treating physician, the patient is no longer benefiting from the treatment, vorasidenib is approved and available by prescription, or the study is terminated.

Requests by treating physicians to file a single patient investigational new drug application as part of the expanded access program for vorasidenib will be considered on a case-by-case basis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females; ages ≥ 12 years old.
2. IDH-mutant oligodendroglioma or astrocytoma with the IDH1 or IDH2 gene mutation confirmed by tissue-based diagnosis.
3. At least 1 prior surgery for glioma (including biopsy).
4. Adequate bone marrow function as evidenced by:

   * Absolute neutrophil count ≥ 1.5 X 109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥ 100 X 109/L
5. Adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN)
   * Aspartate aminotransferase and alanine aminotransferase: at or below the ULN
   * Alkaline phosphatase ≤ 2.5 X ULN
6. Adequate renal function as evidenced by a creatinine clearance (CrCl) ≥ 40 mL/min

   Exclusion criteria:
7. Patient is eligible for a clinical trial with vorasidenib.
8. Patients who are enrolled in a Servier-sponsored clinical trial and have completed all requirements of the trial may be eligible if the patient continues to benefit from vorasidenib and does not meet criteria for discontinuation of treatment.
9. Pregnant or breastfeeding.
10. Patients who require or who cannot withhold strong inhibitors of CYP1A2 (ciprofloxacin and fluvoxamine). Consider alternative therapies that are not strong CYP1A2 inhibitors.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dewey, MD, Study Director — Servier Pharmaceuticals, LLC